CLINICAL TRIAL: NCT05977465
Title: Clinical Study to Investigate the Possible Effect of Empagliflozin in Treatment of Peripheral Diabetic Neuropathy in Patients With Diabetes Mellitus Type 2
Brief Title: Empagliflozin in Treatment of Peripheral Diabetic Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Maha Khalifa, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35200/1/22
Record Dates: First submitted 2023-07-16; First posted 2023-08-04 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Neuropathy Peripheral
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): include twenty-five patients who will receive placebo tablets once daily for three months, plus their antidiabetic drugs ( Dpp4 inhibitor and metformin)
- Empagliflozin group (Experimental): include twenty five patients who will receive Empagloflozin 25 mg once daily for three months, plus their antidiabetic drugs ( Dpp4 inhibitor and metformin)
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — treatment
  Other Names: empagliflozin tablets
  Arms: Empagliflozin group

SUMMARY:
The aim of the study is to investigate the possible protective effect of empagliflozin in patients with type 2 diabetes mellitus with diabetic peripheral neuropathy and not on SGLT2 inhibitors treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes mellitus (Hba1c 7 %- 9%). Patients receiving dipeptidyl peptidase-4 inhibitors, metformin ± basal insulin.

Patients with peripheral neuropathy and not on SGLT2 inhibitor treatment. Patients aged between 18 years old to 65 years old.

Exclusion Criteria:

* Breastfeeding female.
* Pregnant female.
* Estimated Glomerular Filtration Rate less than 45 mL/minute/1.73 m2.
* Patients with type 1 diabetes mellitus.
* Patients with diabetic ketoacidosis.
* Patients with urinary tract infections.
* Dehydrated patients till normalized.
* Lower limb amputation patients.
* SGLT2 inhibitors hypersensitivity.
* Severe hepatic patients.
* Patients on neuroprotective drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Change in the electrophysiological assessment of sensory and motor nerve conduction of the lower limb extremities. | change from baseline at three month
  The electrophysiological studies will be performed using Nihon Kohden Neuropack, six-channel apparatus (Nihon Kohden, Japan) using surface electrodes, for the two studied groups.
Change in HbA1c % | change from baseline at three months
  HbA1c % will be assayed in whole blood using an automated System (H.P.L.C model: G89051, Tosoh, USA), for the two studied groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Khalifa, Pharm D, Principal Investigator — Tanta University
Locations (1):
- Faculty of pharmacy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] El-Haggar SM, Hafez YM, El Sharkawy AM, Khalifa M. Effect of empagliflozin in peripheral diabetic neuropathy of patients with type 2 diabetes mellitus. Med Clin (Barc). 2024 Jul 26;163(2):53-61. doi: 10.1016/j.medcli.2024.01.027. Epub 2024 Apr 22. English, Spanish. PMID 38653618